CLINICAL TRIAL: NCT03329248
Title: NANT Pancreatic Cancer Vaccine: Molecularly Informed Integrated Immunotherapy Combining Innate High-affinity Natural Killer (haNK) Cell Therapy With Adaptive T-cell Therapy (Adenovirus, Yeast, Fusion Protein Vaccine) in Subjects With Pancreatic Cancer Who Have Progressed on or After Standard-of-care Therapy
Brief Title: QUILT-3.060: NANT Pancreatic Cancer Vaccine: Molecularly Informed Integrated Immunotherapy in Subjects With Pancreatic Cancer Who Have Progressed on or After Standard-of-care Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.060
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ALT-803; avelumab; Bevacizumab; Capecitabine; Cyclophosphamide; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Omacor; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NANT Pancreatic Cancer Vaccine (Experimental): A combination of agents will be administered to subjects in this study: ALT-803, ETBX-011, GI-4000, haNK, avelumab, bevacizumab, capecitabine, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, omega-3-acid ethyl esters, oxaliplatin, SBRT
  Interventions: Biological: ALT-803; Biological: ETBX-011; Biological: GI-4000; Biological: haNK for infusion; Biological: avelumab; Biological: bevacizumab; Drug: Capecitabine; Drug: Cyclophosphamide; Drug: Fluorouracil; Drug: Leucovorin; Drug: nab-Paclitaxel; Drug: lovaza; Drug: Oxaliplatin; Procedure: SBRT

INTERVENTIONS:
Biological: ALT-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
Biological: GI-4000 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins
Biological: haNK for infusion — NK-92 [CD16.158V, ER IL-2]
Biological: avelumab — Recombinant human anti-PD-L1 IgG1 monoclonal antibody
Biological: bevacizumab — Recombinant human anti-VEGF IgG1 monoclonal
Drug: Capecitabine — 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
Drug: Leucovorin — L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
Drug: nab-Paclitaxel — Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
Drug: lovaza — Omega-3-acid ethyl esters
Drug: Oxaliplatin — cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum
Procedure: SBRT — Stereotactic Body Radiation Therapy

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of metronomic combination therapy in subjects with pancreatic cancer who have progressed on or after previous SoC chemotherapy. Phase 2 will be based on Simon's two-stage optimal design.

DETAILED DESCRIPTION:
Treatment will be administered in two phases, an induction and a maintenance phase, as described below. Subjects will continue induction treatment for up to 1 year. Treatment in the study will be discontinued if the subject experiences progressive disease (PD) or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. Those who have a complete response (CR) in the induction phase will enter the maintenance phase of the study. Subjects may remain on the maintenance phase of the study for up to 1 year. Treatment will continue in the maintenance phase until the subject experiences PD or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. The maximum time on study treatment, including both the induction and maintenance phases, is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically-confirmed pancreatic cancer with progression on or after SoC therapy.
4. ECOG performance status of 0 to 2.
5. Have at least 1 measurable lesion of ≥ 1.5 cm.
6. Must have a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen following the conclusion of the most recent anticancer treatment and be willing to release the specimen. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide blood samples prior to the start of treatment on this study.
8. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment, if considered safe by the Investigator.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. History of persistent grade 2 or higher (CTCAE Version 4.03) hematological toxicity resulting from previous therapy.
2. Within 5 years prior to first dose of study treatment, any evidence of other active malignancies or brain metastasis except controlled basal cell carcinoma; prior history of in situ cancer (eg, breast, melanoma, cervical); prior history of prostate cancer that is not under active systemic treatment (except hormonal therapy) and with undetectable prostate-specific antigen (PSA) (< 0.2 ng/mL); bulky (≥ 1.5 cm) disease with metastasis in the central hilar area of the chest and involving the pulmonary vasculature.
3. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
4. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
5. History of organ transplant requiring immunosuppression.
6. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
7. Requires whole blood transfusion to meet eligibility criteria.
8. Inadequate organ function, evidenced by the following laboratory results:

   1. White blood cell (WBC) count < 3,500 cells/mm3
   2. Absolute neutrophil count < 1,500 cells/mm3.
   3. Platelet count < 100,000 cells/mm3.
   4. Hemoglobin < 9 g/dL.
   5. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   6. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   7. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   8. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
9. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
10. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
11. Positive results of screening test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
12. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
13. Known hypersensitivity to any component of the study medication(s).
14. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
15. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
16. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
17. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
18. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
19. Concurrent participation in any interventional clinical trial.
20. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 1b portion of the study enrolled participants. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study.
  Eligible participants could have gone through both induction and maintenance treatment on study.
Groups:
- NANT Pancreatic Cancer Vaccine: A combination of agents were administered to subjects in this study: ALT-803, ETBX-011, GI-4000, haNK, avelumab, bevacizumab, capecitabine, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, omega-3-acid ethyl esters, oxaliplatin, SBRT ALT-803: Recombinant human super agonist interleukin-15 (IL-15) complex ETBX-011: Ad5 [E1-, E2b-]-CEA GI-4000: Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins haNK for infusion: NK-92 [CD16.158V, ER IL-2] avelumab: Recombinant human anti-PD-L1 IgG1 monoclonal antibody bevacizumab: Recombinant human anti-VEGF IgG1 monoclonal Capecitabine: 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine Cyclophosphamide: 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate Fluorouracil: 5-fluoro-2,4 (1H,3H)-pyrimidinedione Leucovorin: L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt nab-Paclitaxel: Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin lovaza: Omega-3-acid ethyl esters Oxaliplatin: cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum SBRT: Stereotactic Body Radiation Therapy
Period: Overall Study
Arm/Group | NANT Pancreatic Cancer Vaccine
Started | 6
Completed | 0
Not Completed | 6
Not completed — Progressive Disease | 6

BASELINE CHARACTERISTICS:
Groups:
- NANT Pancreatic Cancer Vaccine: A combination of agents will be administered to subjects in this study: ALT-803, ETBX-011, GI-4000, haNK, avelumab, bevacizumab, capecitabine, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, omega-3-acid ethyl esters, oxaliplatin, SBRT ALT-803: Recombinant human super agonist interleukin-15 (IL-15) complex ETBX-011: Ad5 [E1-, E2b-]-CEA GI-4000: Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins haNK for infusion: NK-92 [CD16.158V, ER IL-2] avelumab: Recombinant human anti-PD-L1 IgG1 monoclonal antibody bevacizumab: Recombinant human anti-VEGF IgG1 monoclonal Capecitabine: 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine Cyclophosphamide: 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate Fluorouracil: 5-fluoro-2,4 (1H,3H)-pyrimidinedione Leucovorin: L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt nab-Paclitaxel: Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin lovaza: Omega-3-acid ethyl esters Oxaliplatin: cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum SBRT: Stereotactic Body Radiation Therapy
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Subjects with pancreatic cancer who have progressed on or after previous SoC chemotherapy [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: Graded Using the National Cancer Institute(NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Time Frame: 30 days after last dose, up to 2 years (up to 1 year in each treatment phase) or until they experience confirmed progressive disease or unacceptable toxicity, withdrawn consent, or if the Investigator feels it is no longer in their best interest.
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Participants
  Treatment Emergent Adverse Events | 6
  Treatment Emergent Serious Adverse Events | 3

2. Secondary Outcome: Objective Response Rate by RECIST Version 1.1
Time Frame: Tumors will be assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression, up to 211 days.
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Objective Response Rate by irRC
Time Frame: Tumors will be assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until confirmed disease progression, up to 211 days.
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Progression Free Survival by RECIST Version 1.1.
Time Frame: Tumors will be assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression or death
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Months | 4.8 [1.9 to NA] — Not Achieved

5. Secondary Outcome: Progression Free Survival by irRC
Time Frame: Tumors will be assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until confirmed disease progression or death
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Months | 4.8 [1.9 to NA] — Not Achieved

6. Secondary Outcome: Overall Survival
Time Frame: Tumors will be assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until death
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Months | 7.3 [5.0 to NA] — Not Achieved

7. Secondary Outcome: Duration of Response (DOR) by RECIST Version 1.1 and irRC
Description: DOR was be defined as the time from the date of first response (PR or CR) to the date of disease progression or death (any cause) whichever occurs first. Responding subjects completed study follow-up or initiating a new anticancer therapy prior to documented PD were censored in the DOR analysis at the last known date the subject was progression free prior completing follow-up or initiating the new therapy.
Time Frame: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until confirmed disease progression, up to 211 days
Population: There were no participants with confirmed CR or PR. Therefore, no participants were included in the DOR analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Months | NA [NA to NA] — Insufficient number of participants with events.

8. Secondary Outcome: Disease Control Rate (Confirmed Complete Response, Partial Response, or Stable Disease Lasting for at Least 2 Months) by RECIST Version 1.1.
Description: Disease control is defined as subjects with a confirmed CR, PR, or SD lasting for at least 2 months.
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Participants
  Confirmed Complete Response | 0
  Confirmed Partial Response | 0
  Unconfirmed Complete Response | 0
  Unconfirmed Partial Response | 0
  Stable Disease | 5
  Progressive Disease | 1

9. Secondary Outcome: Quality of Life by Patient Reported Outcomes (PRO)
Description: PROs were assessed using the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaire. The FACT-Hep is compilation of general questions divided into five QOL subscales:
  Physical Well-Being - Scores ranging from 0-28 Social/Family Well-Being - Scores ranging from 0-28 Emotional Well-Being - Scores ranging from 0-24 Functional Well-Being - Scores ranging from 0-28 Additional Concerns - Scores ranging from 0-72 It uses 5-point Likert-type response categories ranging from 0 = 'not at all' to 4 = 'very much'.
  The higher scales and subscales indicate better quality of life. Negatively worded items were reverse scored. If the missing for each subscale was less than 50%, the prorating scores were computed for the subscale.
Time Frame: Up to 9 months
Population: Not all participants had QOLs collected for analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
score on a scale
  Additional Concerns - Baseline: number analyzed (Participants) | 5
  Additional Concerns - Baseline | 44.0 [39.0 to 65.0]
  Emotional Well-Being - Baseline: number analyzed (Participants) | 5
  Emotional Well-Being - Baseline | 14.0 [12.0 to 21.0]
  Functional Well-Being - Baseline: number analyzed (Participants) | 5
  Functional Well-Being - Baseline | 19.0 [13.0 to 23.0]
  Physical Well-Being - Baseline: number analyzed (Participants) | 5
  Physical Well-Being - Baseline | 16.0 [10.0 to 25.0]
  Social/Family Well-Being - Baseline: number analyzed (Participants) | 5
  Social/Family Well-Being - Baseline | 25.0 [18.7 to 28.0]
  Additional Concerns - End of Dosing: number analyzed (Participants) | 5
  Additional Concerns - End of Dosing | 46.0 [27.0 to 55.0]
  Emotional Well-Being - End of Dosing | 12.5 [9.0 to 22.0]
  Functional Well-Being - End of Dosing | 13.0 [8.0 to 22.0]
  Physical Well-Being - End of Dosing | 15.0 [5.0 to 26.0]
  Social/Family Well-Being - End of Dosing | 22.6 [13.0 to 28.0]

10. Secondary Outcome: Disease Control Rate (Confirmed Complete Response, Partial Response, or Stable Disease Lasting for at Least 2 Months) by irRC
Description: Disease control is defined as subjects with a confirmed CR, PR, or SD lasting for at least 2 months.
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 6
Participants
  Confirmed irCR | 0
  Confirmed irPR | 0
  Unconfirmed irCR | 0
  Unconfirmed irPR | 0
  irSD | 4
  Unconfirmed irPD | 0
  Confirmed irPD | 2

ADVERSE EVENTS:
Time Frame: Non-serious AEs were followed for 30 days after the subject's last dose of study treatment, up to 2 years. Non-serious grade 3 or 4 AEs were followed until resolution or stabilization, up to 2 years. All SAEs that had not resolved upon discontinuation of the subject's participation in the study were followed until recovered, recovered with sequelae, not recovered (death due to other cause), death (due to the SAE), lost to follow-up.
Arm/Group | NANT Pancreatic Cancer Vaccine
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Pancreatic Cancer Vaccine (N=6)
Abdominal pain (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Obstruction gastric (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Abdominal abscess (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Pancreatic Cancer Vaccine (N=6)
Neutropenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Injection site reaction (General disorders) | 6
Pyrexia (General disorders) | 5
Injection site erythema (General disorders) | 4
Injection site pain (General disorders) | 4
Chills (General disorders) | 3
Injection site swelling (General disorders) | 3
Asthenia (General disorders) | 2
Disease progression (General disorders) | 2
Influenza like illness (General disorders) | 2
Mucosal inflammation (General disorders) | 2
Catheter site irritation (General disorders) | 1
Chest pain (General disorders) | 1
Feeling abnormal (General disorders) | 1
Injection site bruising (General disorders) | 1
Injection site oedema (General disorders) | 1
Injection site pruritus (General disorders) | 1
Injection site warmth (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 5
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Renal injury (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Labile blood pressure (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3
Procedural pain (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Vulvovaginal injury (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Tachycardia (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Diplopia (Eye disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Breast pain (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT03329248/Prot_SAP_000.pdf